CLINICAL TRIAL: NCT04322409
Title: The Role of Neuromuscular Electrical Stimulation (NMES) on Improving Function in Individuals With Chronic Ankle Instability
Brief Title: NMES and Chronic Ankle Instability
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Appalachian State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 20-042
Record Dates: First submitted 2020-01-07; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Chronic Ankle Instability
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: 2x3 Factorial; 2 groups by 3 time points
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NMES (Experimental): The experimental treatment of Neuromuscular Electrical Stimulation over the Peroneus Longus.
  Interventions: Device: Neuromuscular Electrical Stimulation
- TENS (Placebo Comparator): The placebo treatment of Transcutaneous Electrical Nerve Stimulation over the same region as the peroneus longus
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — 5 sessions that consist of NMES over the peroneus longus muscle. This consists of a biphasic current with a phase duration of 240us delivered in a frequency of 75 pules per second, with a ramp-up time of 2-seconds, followed by a 50-s rest period (no stimulation). Each cycle will consist of 10 seconds of "on" time, and 50 seconds off, with 10 cycles being performed each session.
  Other Names: NMES
  Arms: NMES
Device: Transcutaneous Electrical Nerve Stimulation — 5 sessions that consist of 11-minutes of TENS over the skin of the peroneus longus. This consists of a biphasic current will be continuously applied at 100 pulses per second, with a phase duration of 100us for 10 minutes. The intensity will be turned up until the point the subjects feel the current (sensory threshold)
  Other Names: TENS
  Arms: TENS

SUMMARY:
Chronic ankle instability is associated with changes in the nervous system that amount to increased difficulty in activating the stabilizing muscles of the ankle. Neuromuscular Electrical Stimulation involves using electricity to activate those muscles in bursts, and is commonly used to improve muscle function in those with ACL injury. This study will provide 5 treatments over 2 weeks in patients with Chronic Ankle Instability and determine if Electrical Stimulation can change neural excitability, balance, neuromuscular control, and perceived function in these individuals.

DETAILED DESCRIPTION:
Individuals with joint injuries, including ankle sprain and anterior cruciate ligament (ACL) injury have been observed to exhibit changes in central nervous system function that potentially predispose them for further injury (Needle et al. 2017). In ankle sprains, repeated sensations of rolling and giving-way known as chronic ankle instability (CAI) emerges in nearly 50 percent of those with a history of ankle sprain (Holland et al. 2019), with symptoms tied to changes in central nervous system function. As the understanding of these pathologies have expanded, researchers have begun to attempt to identify neuromodulatory interventions capable of addressing injury-induced maladaptive neuroplasticity, thus improving function (Bruce et al. 2020, In Press).

Among those with ACL injury, one of the most common interventions implemented to overcome muscle activation deficits includes neuromuscular electrical stimulation (NMES) (Lepley et al. 2015). This intervention is often used in the initial stages of post-surgical recovery to improve quadriceps function; however, it's use in other populations of joint injury (i.e. ankle sprain) is far more limited. Some previous research has looked at the effects of NMES on acute ankle sprains, as this is the timeframe in which muscle activation deficits would be most evident (Wainwright et al. 2019), but there is very limited evidence in those with CAI. It was potentially thought that activation deficits are less evident and strengthening may overcome these deficits in those with chronic injury; however, new insights have identified additional mechanisms by which NMES may be effective (Lepley et al. 2015). Aside from generating activation of a generally inactive muscle, NMES when performed at high intensities has been described to improve neuromuscular function through disinhibitory mechanisms. That is that increased somatosensation from the electrical stimulation raises the central nervous sytem's awareness of that muscle's activation, yielding decreased inhibition and ultimately increased neural excitability.

Our previous research using cortically-directed interventions demonstrated that improving neural excitability yielded better function in patients with chronic ankle instability (Bruce et al. 2020). This study will follow a similar framework; however, determining if these changes can be induced via a peripheral intervention. These findings have the ability to reframe the current treatment for CAI.

We are pursuing the following 2 specific aims:

1. To determine if NMES changes neural excitability (MEP size, H:M ratio, silent period) compared to a placebo treatment in participants with chronic ankle instability.

   H1: NMES will increase MEP size, H:M ratio, and decrease cortical silent period in individuals with CAI compared to the placebo treatment.
2. To determine if changes in neural excitability related to NMES or placebo treatment result in improved function (balance, muscle activation, outcomes) in participants with chronic ankle instability.

H2: Increased neural excitability will yield improved balance (postural stability indices), muscle activation, and patient-reported function.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be healthy subjects between the ages of 18-35. The primary inclusion criteria for this study is the presence of chronic ankle instability (CAI). According to guidelines from the International Ankle Consortium, this means subjects will report having a history of one or more ankle sprains (the first >1 year ago), and repeated sensations of giving-way as measured by a score >10 on the Identification of Functional Ankle Instability instrument (IDFAI).

Exclusion Criteria:

* History of fracture or surgery to the legs
* Injury to the lower legs within 3 months prior to reporting for testing that resulted in modified physical activity.
* Currently involved in an ankle rehabilitation program.
* Failing to meet standards for the safe practice of transcranial magnetic stimulation and transcranial direct current stimulation (See questionnaire). Briefly, this includes personal or family history of seizure or epilepsy; current medication use that raises risk of seizure; implanted metal, medication devices, etc.; history of brain or heart surgery; and sensitivity of the scalp or skin.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Tibialis Anterior corticospinal excitability | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Motor evoked potential size of tibialis anterior
Soleus corticospinal excitability | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Motor evoked potential size of soleus
Peroneus Longus corticospinal excitability | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Motor evoked potential size of peroneus longus
Tibialis anterior reflexive excitability | Baseline, Week-2 (end of intervention), Week-4 (retention)
  H:M ratio of tibialis anterior
Soleus reflexive excitability | Baseline, Week-2 (end of intervention), Week-4 (retention)
  H:M ratio of soleus
Peroneus longus reflexive excitability | Baseline, Week-2 (end of intervention), Week-4 (retention)
  H:M ratio of peroneus longus

SECONDARY OUTCOMES:
Dynamic postural stability index | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Postural stability indices during a hop-to-stabilization task
Tibialis Anterior muscle activation | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Mean electromyography from the tibialis anterior during a hop-to-stabilization task
Soleus muscle activation | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Mean electromyography from the soleus during a hop-to-stabilization task
Peroneus Longus muscle activation | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Mean electromyography from the peroneus during a hop-to-stabilization task
Ankle Eversion Strength | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Isometric ankle eversion strength
Side-to-side Hop Test | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Time to complete 10 hops over 30 cm lines
Patient-reported outcomes | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Foot & Ankle ability measure, Disablement in the Physically Active Scale, Tampa Scale for Kinesiophobia
Foot & Ankle ability measure | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Subjects complete FAAM questionnaire
Disablement in the Physically Active Scale | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Subjects complete DPA questionnaire
Tampa Scale for Kinesiophobia | Baseline, Week-2 (end of intervention), Week-4 (retention)
  Subjects complete TSK-11 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Leon Levine Hall for Health Sciences, Boone, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Needle AR, Tinsley JE, Cash JJ, Koeval BK, Barton JA, Howard JS. The effects of neuromuscular electrical stimulation to the ankle pronators on neural excitability & functional status in patients with chronic ankle instability. Phys Ther Sport. 2023 Mar;60:1-8. doi: 10.1016/j.ptsp.2022.12.001. Epub 2022 Dec 9. PMID 36634453